CLINICAL TRIAL: NCT05859126
Title: The Effect of Maternal Choline Supplementation on Offspring Cognition in Adolescence: A 13 Year Follow-up of a Randomized Feeding Study
Brief Title: Maternal Choline Supplementation and Offspring Cognition in Adolescence
Acronym: CholTeens
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB0147236
Record Dates: First submitted 2023-03-30; First posted 2023-05-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Deficit in Attention; Executive Dysfunction; Emotional Regulation
Keywords: adolescence; emotion; cognition; choline
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Choline Supplementation 930 mg/d (Experimental): Supplementation of 930 mg/d from early second trimester through birth. Offspring are followed for cognitive outcomes.
  Interventions: Dietary Supplement: Maternal Choline Supplementation 930 mg/d
- Maternal Choline Supplementation 480mg/d (Active Comparator): Supplementation of 480 mg/d from early second trimester through birth.Offspring are followed for cognitive outcomes.
  Interventions: Dietary Supplement: Maternal Choline Supplementation 480 mg/d

INTERVENTIONS:
Dietary Supplement: Maternal Choline Supplementation 930 mg/d — Mothers were supplemented with choline (930mg/d) from second trimester through birth. This is a 13 year follow up of their offspring.
  Arms: Maternal Choline Supplementation 930 mg/d
Dietary Supplement: Maternal Choline Supplementation 480 mg/d — Mothers were supplemented with choline (480 mg/d) from second trimester through birth. This is a 13 year follow up of their offspring.
  Arms: Maternal Choline Supplementation 480mg/d

SUMMARY:
The goal of this 13-year follow up of a randomized control trial is to study the effect of maternal choline supplementation on offspring cognition in adolescence.

The main question[s] it aims to answer are:

Does a higher dose of maternal choline choline (930 mg/d day supplementation) lead to improved cognition in adolescence including hippocampal-dependent episodic memory and executive functioning when compared to lower dose supplementation (480 mg/d).

In this follow-up of a clinical trial participants will complete online cognition testing and emotion testing.

DETAILED DESCRIPTION:
Eggs are one of the richest dietary sources of choline, an essential nutrient that plays critical roles in fetal development, including shaping the structure and function of the offspring brain. Furthermore, evidence shows that pregnancy dramatically increases the demand for choline.

In rodents consuming standard chow, pregnancy results in a pronounced depletion of maternal choline pools, indicating that choline requirements during pregnancy are increased and that maternal and fetal requirements likely exceed the amount typically consumed by mothers. Additionally, human research from the investigators' laboratory has found that the "Adequate Intake" (AI) levels for choline during pregnancy, set in 1998 and based on the amount needed to prevent liver damage in adult men, may not be sufficient to meet the demands of pregnancy. Specifically, pregnant women consuming choline at the AI level have significantly lower circulating concentrations of several choline metabolites compared to non-pregnant women, and even doubling maternal choline intake (to twice the AI) fails to produce the metabolite levels observed in non-pregnant women. Perhaps most importantly, a substantial body of experimental research in animal models demonstrates that supplementation with additional choline during pregnancy significantly improves lifelong memory, attention, and emotional regulation in offspring, re-duces or eliminates normal ageing-related decline in cognitive function, and reduces the im-pact of a range of prenatal neural insults (e.g., alcohol exposure, maternal stress).

Despite extensive experimental data in animal models demonstrating lasting beneficial effects of maternal choline supplementation on offspring memory, attention, and affect, few studies have evaluated the effects of increasing maternal choline intake in humans. Moreover, results from existing human studies are not sufficiently conclusive to alter dietary intake recommendations for pregnancy. However, a randomized choline feeding trial from the investigators' laboratory demonstrated beneficial effects of increased maternal choline intake (930 mg/d vs. 480 mg/d) on offspring cognitive functioning during infancy and at 7 years of age (work supported in part by previous ENC funding). Based on these findings, the investigators propose to follow up children born to mothers participating in this trial, to examine longer-term effects of maternal choline supple-mentation on child cognition and emotional well-being at thirteen years of age. This will be the first randomized controlled trial (RCT) following children into adolescence, a time when tests are highly predictive of adult functioning.

Choline is an essential nutrient that plays critical roles in fetal neurodevelopment. The demand for choline increases markedly during pregnancy, indicated by a pronounced depletion of maternal choline pools even when women consume the Adequate Intake (AI) level. It is a concern that fewer than 10% of reproductive age women achieve the recommended AI level, and that choline is not included in standard prenatal vitamin regimens.

Decades of rodent studies show that maternal choline intake affects offspring brain structure, neural function and cognitive performance throughout life the lifespan. Maternal choline deficiency produces lasting offspring cognitive impairment, whereas increasing maternal choline intake markedly improves offspring cognition and provides widespread neuroprotection in various diseases and early insults.

Only 3 Randomized Controlled Trials (RCTs) have evaluated offspring cognition following maternal choline supplementation (MCS) in healthy human pregnancies. One trial conducted in the investigators' lab demonstrated that MCS improves offspring cognition during infancy and early childhood, but no studies have yet determined whether the beneficial effects observed in the immature human brain are maintained in adulthood. This question can be addressed by assessing the cognitive performance of MCS offspring in adolescence, a time when many neurocognitive tests are strong predictors of ultimate adult functioning.

The planned study will take advantage of the unique opportunity to follow up the offspring of women who participated in a controlled feeding study comparing two levels of choline intake during pregnancy: 480 vs 930 mg/d. The offspring will be tested at 13 years old, an age when cognitive functioning predicts adult functioning. The investigators predict that the cognitive performance of the children born to women consuming 480 mg/d (approximately the AI) during the last trimester of pregnancy will be poorer than children born to women consuming 930 mg/d.

The predicted results would strongly indicate that the low choline intake of most pregnant women impedes the lifelong cognitive functioning of their children. Demonstrating this effect would spur the addition of choline to standard prenatal vitamin regimens-the predicted result being population-wide improvements in cognitive functioning, in part due to widespread neuroprotection. These effects would be particularly beneficial for at-risk pregnancies and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of mothers from the original choline feeding trial
* Testing will commence when the child reaches 13 years of age (determined by date of birth of participant)

Exclusion Criteria:

* Failure to follow the study protocol regarding test procedures and questionnaires
* Lack of internet access with the requisite speed and stability needed to support the online testing tools

Ages: 13 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
CANTAB Signal Detection test | at 13 years of age
  To measure selective and sustained attention where sensitivity to stimulus ranges from 0 (bad) to 1 (good)
CANTAB Delayed Matching to Sample | at 13 years of age
  To measure memory where scoring is based on percent correct where 0% is bad and 100% is excellent), Paired Associates Learning (where scoring is based on total errors, where 0 is best), and Pattern Recognition Memory (where outcome is measured as percentage of correct trials and latency (speed of participant's response).)
CANTAB Spatial Working Memory | at 13 years of age
  To measure executive function (where outcome measure is number of errors and lower is better),
CANTAB Cambridge Gambling | at 13 years of age
  To measure executive function (where outcome measure is number of errors and lower is better),

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) | at 13 years of age
  To measure emotion regulation where scoring is from 0-226 and lower is better.
Youth Self Report (CBCL | at 13 years of age
  To measure emotion regulation where scoring is from 0-226 and lower is better.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Strupp, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Division of Nutritional Sciences, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth SA, Lam AE, Strupp BJ, Canfield RL, Larson EA. The Effect of Maternal Choline Intake on Offspring Cognition in Adolescence: Protocol for a 14-year Follow-Up of a Randomized Controlled Feeding Trial. JMIR Res Protoc. 2025 Jul 11;14:e73508. doi: 10.2196/73508. PMID 40644695

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05859126/SAP_000.pdf